CLINICAL TRIAL: NCT03564756
Title: Effect of Ascorbic Acid Supplementation in Pregnancy on Anemia (AAA)
Acronym: AAA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty with enrollment
Sponsor: Fetal Medicine Foundation (Other)
Collaborators: Wright State University (Other); Five Rivers Health Centers (Unknown)
Responsible Party: Principal Investigator, David S. McKenna, Principal Investigator, Fetal Medicine Foundation
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AAA-001
Record Dates: First submitted 2018-05-25; First posted 2018-06-21 (Actual); Last update posted 2022-09-22 (Actual); Status verified 2022-09

CONDITIONS: Anemia in Pregnancy
Keywords: Anemia; Pregnancy; Iron; Vitamin C
MeSH Terms: conditions — Anemia | interventions — Ascorbic Acid

STUDY DESIGN:
Intervention Model Description: Randomized Parallel Group, Placebo Controlled Trial
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Iron + Vitamin C (Experimental): One iron tablet once a day plus a 500 mg vitamin C tablet twice a day until delivery.
  Interventions: Dietary Supplement: Vitamin C
- Iron + Placebo (No Intervention): One iron tablet once a day plus a placebo tablet twice a day until delivery.

INTERVENTIONS:
Dietary Supplement: Vitamin C — 1000mg Vitamin C per day
  Other Names: Ascorbic Acid
  Arms: Iron + Vitamin C

SUMMARY:
A. Anemia is a common problem affecting pregnancy and can result in profound consequences to both the mother and the growing fetus. Current treatment usually includes administration of oral or IV iron, or blood transfusions. Vitamin C is known to affect iron metabolism and has been shown to improve outcomes when used in addition to iron, however, few studies have been performed in pregnancy. The primary aim of this study is to identify the effects of vitamin C on anemia in pregnancy. The Investigators propose a double-blind, randomized placebo controlled trial of 1000mg vitamin C supplementation in 200 low risk pregnancies with iron-deficiency anemia. All newly enrolled patients, who meet inclusion and exclusion criteria, will receive the standard of care evaluation and treatment for anemia in pregnancy. Additionally, patients will be randomized to receive either placebo or vitamin C and compliance monitored with a pill diary. Data will be analyzed by T tests and Mann-Whitney U test. If the data shows a positive statistical significance, vitamin C may be a useful supplement to iron in treating anemia.

DETAILED DESCRIPTION:
A. Anemia is the most common hematological abnormality during pregnancy and was found to affect 24.1% of pregnant women in a WHO study.2 The most common types of anemia affecting pregnancy are iron-deficiency and acute blood loss. Vitamin C, also known as ascorbic acid, has been well documented to play an active role in the absorption and metabolism of iron from the gut.6 Vitamin C has been used in studies to treat anemic non-pregnant women resulting in significant increases in hemoglobin levels. Similar effects have been found in multiple studies using vitamin C as adjunct treatment for hemodialysis patients with non-responsive anemia.10,12 Vitamin C has already been extensively studied in pregnant women for its effects on preeclampsia, preterm birth, neonatal morbidity and other outcomes, and found to have no adverse effects in doses as high as 1000mg daily or in combination with other medications.8 After an extensive literature search, very few studies have been performed assessing the effect on hemoglobin levels after vitamin C supplementation. One study by Sharma et al. supplemented pregnant women with 500mg vitamin C and found a 18.04% increase in hemoglobin compared to 5.49% in the control.11 A Cochran Review of 29 studies did not discuss or evaluate the effects of vitamin C on anemia.8 Due to the minimal side-effect profile and potential benefits of successfully treating anemia, further research in the area is needed.

V. SPECIFIC AIMS OR OBJECTIVES A. To perform a double-blinded, randomized placebo controlled trial of 1000mg vitamin c supplementation on iron-deficiency anemia in low-risk pregnancies.

VI. SIGNIFICANCE TO PATIENT, INSTITUTION, PROFESSION, OR ALL A. Anemia has been associated with adverse maternal and fetal outcomes, to include, but not limited to low birth weight, preterm delivery, perinatal mortality and postpartum depression.1 Per ACOG guidelines, all pregnant women should be screened for anemia, evaluated for causes and provided supplemental iron. A study by Sharma et al has already demonstrated a significant increase in hemoglobin levels in pregnancy with 500mg vitamin C supplementation.11 Due to the paucity of research of vitamin C in pregnancy, further studies are needed to determine reproducibility.

VII. METHODS A. The investigators plan to enroll 200 patients total, 100 per arm. Potential subjects will be screened by study personal from the new intakes for prenatal care in the Five Rivers Center for Women's Health. A complete blood count (CBC) is obtained as standard of care at the first prenatal visit. The CBC includes hemoglobin level, hematocrit, and red blood cell indices (i.e. MCV and MCH). Pregnant women in the first half of their pregnancy who are found to have a hematocrit level less than 33% (Caucasian and other races), and less than 31% (African American women), will be potentially eligible for enrollment. Women who are noted to be anemic per these thresholds will have iron studies (iron, transferrin, ferritin) and hemoglobin electrophoresis (if not already performed), as part of the standard of care for the evaluation of anemia during pregnancy.1 Inclusion criteria consists of gestational age at enrollment less than 20 0/7 weeks, singleton gestation, iron deficiency anemia defined as maternal serum ferritin levels less than 15 micrograms/dL, and planned delivery at Miami Valley Hospital. Exclusion criteria consist of vitamin C use >150mg/day (typical prenatal vitamin contains 60mg Vitamin C), diabetes (gestational, types 1,2); chronic medical disease; known or discovered hemoglobinopathy (including heterozygous states); known metabolic disease that may contribute to impaired iron absorption (including a history of bariatric surgery, renal disease and an inability to tolerate oral iron); known fetal abnormalities; participation in another interventional trial; illicit drug or alcohol use. All risks/benefits will be reviewed and all questions answered prior to the patient being enrolled. Written informed consent will be obtained by a study investigator or qualified personnel. Gestational dating will be based upon the best obstetrical estimate.

B. A compounding pharmacy will make 30,000 placebo capsules containing an inert substance (i.e. silica based cellulose), identical appearing to 30,000 capsules of 500mg vitamin C. The pharmacy will package 300 pills of either placebo or vitamin C into 200 boxes, labeled only with the project name and a number. A key containing the known substance of each box and number will be kept by the pharmacy until the end of the study. The boxes will be stored in a secured area of the principal investigators office. The boxes will be taken to Five Rivers Women's Health Clinic to be distributed to enrolled patients. Once enrolled, patients will be given a random box and instructed to take 1 pill twice daily. Patients will be instructed to record pill usage daily for compliance. The patient's name and assigned box number will be kept in a locked cabinet. At the end of the study, the two keys will be compared to determine who received placebo or vitamin C. Both groups will receive prescriptions for ferrous sulfate, 65mg taken once daily; docusate sodium to be taken as needed for constipation; and prenatal vitamins once daily. Patients will receive follow up labs as part of the standard of care for anemia, to include at 28 week, and at delivery. All data will be collected in an Excel spreadsheet, with patient identifiers removed. Data will be analyzed by applying basic T tests and the Mann-Whitney-U test to determine the changes in lab values of hemoglobin, hematocrit, iron, transferrin, ferritin between experimental and control before and after treatment.

ELIGIBILITY:
Inclusion Criteria:

* gestational age at enrollment less than 20 0/7 weeks,
* singleton gestation,
* iron deficiency anemia defined as maternal serum ferritin levels less than 15 micrograms/dL, and
* planned delivery at Miami Valley Hospital.

Exclusion Criteria:

* vitamin C use >150mg/day (typical prenatal vitamin contains 60mg Vitamin C),
* diabetes (gestational, types 1,2); chronic medical disease;
* known or discovered hemoglobinopathy (including heterozygous states);
* known metabolic disease that may contribute to impaired iron absorption (including a history of bariatric surgery, renal disease and an inability to tolerate oral iron);
* known fetal abnormalities;
* participation in another interventional trial;
* illicit drug or alcohol use

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 0 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Change in serum hemoglobin | To be measured at 1st prenatal visit, 28 weeks', and at delivery
  Change in serum hemoglobin

CONTACTS AND LOCATIONS:
Locations (1):
- Five Rivers Health Centers, Dayton, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data will be used by the study team to test the study hypothesis

REFERENCES:
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin No. 95: anemia in pregnancy. Obstet Gynecol. 2008 Jul;112(1):201-7. doi: 10.1097/AOG.0b013e3181809c0d. Erratum In: Obstet Gynecol. 2020 Jan;135(1):222. doi: 10.1097/AOG.0000000000003624. PMID 18591330
- [Background] McLean E, Cogswell M, Egli I, Wojdyla D, de Benoist B. Worldwide prevalence of anaemia, WHO Vitamin and Mineral Nutrition Information System, 1993-2005. Public Health Nutr. 2009 Apr;12(4):444-54. doi: 10.1017/S1368980008002401. Epub 2008 May 23. PMID 18498676
- [Background] Abdel Moety GAF, Ali AM, Fouad R, Ramadan W, Belal DS, Haggag HM. Amino acid chelated iron versus an iron salt in the treatment of iron deficiency anemia with pregnancy: A randomized controlled study. Eur J Obstet Gynecol Reprod Biol. 2017 Mar;210:242-246. doi: 10.1016/j.ejogrb.2017.01.003. Epub 2017 Jan 3. PMID 28073037
- [Background] Hanieh S, Ha TT, Simpson JA, Braat S, Thuy TT, Tran TD, King J, Tuan T, Fisher J, Biggs BA. Effect of low-dose versus higher-dose antenatal iron supplementation on child health outcomes at 36 months of age in Viet Nam: longitudinal follow-up of a cluster randomised controlled trial. BMJ Glob Health. 2017 Sep 22;2(3):e000368. doi: 10.1136/bmjgh-2017-000368. eCollection 2017. PMID 29018582
- [Background] Joseph B, Ramesh N. Weekly dose of Iron-Folate Supplementation with Vitamin-C in the workplace can prevent anaemia in women employees. Pak J Med Sci. 2013 Jan;29(1):47-52. doi: 10.12669/pjms.291.3016. PMID 24353506
- [Background] Lane DJ, Richardson DR. The active role of vitamin C in mammalian iron metabolism: much more than just enhanced iron absorption! Free Radic Biol Med. 2014 Oct;75:69-83. doi: 10.1016/j.freeradbiomed.2014.07.007. Epub 2014 Jul 15. PMID 25048971
- [Background] Rumbold A, Crowther CA. Vitamin C supplementation in pregnancy. Cochrane Database Syst Rev. 2005 Apr 18;(2):CD004072. doi: 10.1002/14651858.CD004072.pub2. PMID 15846696
- [Background] Pena-Rosas JP, De-Regil LM, Gomez Malave H, Flores-Urrutia MC, Dowswell T. Intermittent oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2015 Oct 19;2015(10):CD009997. doi: 10.1002/14651858.CD009997.pub2. PMID 26482110
- [Background] Sedighi O, Makhlough A, Janbabai G, Neemi M. Comparative study of intravenous iron versus intravenous ascorbic Acid for treatment of functional iron deficiency in patients under hemodialysis: a randomized clinical trial. Nephrourol Mon. 2013 Sep;5(4):913-7. doi: 10.5812/numonthly.12038. Epub 2013 Jul 24. PMID 24350091
- [Background] Sultana T, DeVita MV, Michelis MF. Oral vitamin C supplementation reduces erythropoietin requirement in hemodialysis patients with functional iron deficiency. Int Urol Nephrol. 2016 Sep;48(9):1519-24. doi: 10.1007/s11255-016-1309-9. Epub 2016 May 11. PMID 27170339